CLINICAL TRIAL: NCT05841797
Title: Piloting Risk Stratification and Tailored Interventions With Pregnant and Postpartum Women With HIV in Kenya to Prevent Disengagement From Care and Viral Failure
Brief Title: Evaluation of Problem Management Plus in Pregnant Women With HIV in Kenya
Acronym: Tatua
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Alabama at Birmingham (Other); Kenya Medical Research Institute (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 22-1946
Record Dates: First submitted 2023-04-04; First posted 2023-05-03 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV Transmission; Prevention of Mother to Child Transmission; Linkage to care; Retention in care; Community Mentor Mothers; Mobile intervention; Antiretroviral therapy adherence; Infant Health; Maternal CD4/viral loads; Early infant diagnosis; Acceptability of interventions; Vertical transmission; Mental health
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a pilot hybrid type 2 effectiveness-implementation trial in which pregnant women at higher risk for missed visits and treatment failure are randomized to one of three study arms 1:1:1 standard of care, mHealth PM+, or in-person PM+ and followed through 6 months postpartum. Feasibility, acceptability, intervention satisfaction, and preliminary efficacy on mental health and HIV outcomes (combined outcome of continuous viral suppression and engagement in care) will be assessed.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and care providers will not be blinded to study arm, however investigators and analyst will be.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (SOC) (No Intervention): Standard of Care (SOC): For Arm 1 of the pilot trial, SOC will be implemented. SOC for PWLWH in Kenya is carried out according Kenyan National Guidelines and includes integration of antenatal care, HIV care, and HIV-exposed infant follow up within the maternal-child health clinic through 18-24 months postpartum. Provision of ART, HIV education, and adherence counseling is routinely provided. Psychosocial support is provided by either peer educators or lay health workers. WLWH who miss visits are followed up by phone and then traced in the community to encourage return to care.
  PWLWH undergo routine VL testing six months after ART initiation or at confirmation of pregnancy if already on ART. VLs are performed every six months through breastfeeding.
  Women with VL 200 copies/ml undergo enhanced adherence counseling with repeat VL in three months. While routine screening for IPV and depression are recommended per National Guidelines, they are incompletely implemented.
- In-Person Program Management Plus (PM+) (Experimental): For Arm 2, the investigators will implement the adapted PM+ utilizing the complete manual of operations and adaptation lessons learned in the non-clinical trial portion of the study. The investigators will train mentor mothers to serve as PM+ Helpers. In-person sessions will likely be delivered at home. Sessions will continue after the birth if not completed during pregnancy. PM+ Helpers will debrief regularly on the progress of participants with clinically trained supervisors - both for their own psychological well-being and to ensure that participants receive adequate care.
  Interventions: Behavioral: In-Person Program Management Plus (PM+)
- Mobile Program Management Plus (mHealth PM+) (Experimental): For Arm 3, the investigators will implement the adapted PM+ utilizing the complete manual of operations and adaptation lessons learned in the non-clinical trial portion of the study. The investigators will train mentor mothers to serve as PM+ Helpers. In the mHealth delivered version of PM+, PM+ Helpers will conduct PM+ virtually after an initial meeting to create rapport. Sessions will be delivered by either 1) a PM+ Helper- initiated phone call or 2) a participant-initiated call via a call-in help line. Airtime will be provided so that participation will be free of charge. Sessions will continue after the birth if not completed during pregnancy. PM+ Helpers will debrief regularly on the progress of participants with clinically trained supervisors - both for their own psychological well-being and to ensure that participants receive adequate care.
  Interventions: Behavioral: Mobile Program Management Plus (mHealth PM+)

INTERVENTIONS:
Behavioral: In-Person Program Management Plus (PM+) — PM+ sessions conducted in-person by mentor mothers
  Arms: In-Person Program Management Plus (PM+)
Behavioral: Mobile Program Management Plus (mHealth PM+) — PM+ sessions conducted via phone
  Arms: Mobile Program Management Plus (mHealth PM+)

SUMMARY:
This study includes secondary quantitative analysis, qualitative methods, and hybrid type 2 implementation-effectiveness pilot trial. The overall goal of this protocol is to determine whether risk stratification of PWLWH in conjunction with a tailored psychosocial support intervention can optimize health outcomes for the vulnerable women and infants. This study will be conducted in high-volume, low-resource health facilities in Kisumu County, Kenya, which is a priority area for research among WLWH and one of the highest HIV burden counties.

DETAILED DESCRIPTION:
Among pregnant/postpartum women living with HIV (PWLWH) in low resource, high HIV prevalence settings, access to antiretroviral treatment (ART) has increased dramatically and mother-to-child transmission (MTCT) of HIV has decreased substantially, yet successful outcomes are not universal. Despite a 52% decline in new HIV infections among children under five from 2010-2019, recent UNAIDS data indicate global targets were missed by wide margins, with an estimated 160,000 new pediatric HIV infections annually. Sub-optimal retention of PWLWH is a major contributor to new pediatric infections. This study will be conducted in high-volume, low-resource health facilities in Kisumu County, Kenya, which is a priority area for research among WLWH and one of the highest HIV burden counties. As PMTCT programs in sub-Saharan Africa (SSA) aim for the elimination of MTCT in the context of decreased funding, there is need for research geared towards identifying and supporting the most vulnerable PWLWH with tailored interventions that can be implemented using available resources. This study aims to build on a previous study, Mother and Infant Visit Adherence and Treatment Engagement Study (MOTIVATE, R01HD080477), to develop and implement interventions that can promote proper taking of HIV drugs among PWLWH, namely a risk calculator to identify women at high risk for treatment failure and an adapted Problem Management Plus (PM+) intervention specifically geared towards women identified as high risk. Such interventions are critical in order to identify the most vulnerable PWLWH as early as possible to intervene with effective targeted interventions that will help improve maternal and child health outcomes.

ELIGIBILITY:
Inclusion criteria:

* Pregnant woman living with HIV attending an ANC clinic in Kisumu County, on/initiating ART
* At least 15 years of age
* At least 20 weeks estimated gestational age
* At moderate or critical risk of the combined outcome of treatment disengagement or viral failure according to the risk calculator
* Access to a cell phone (for those who share phones, have disclosed their HIV status to whomever individuals share the phone with.

Exclusion Criteria:

* Imminent plans of suicide and severe impairment due to severe mental, neurological or substance use disorders
* Less than 15 years of age
* Less than 20 weeks estimated gestational age or not currently pregnant
* Not HIV-infected at time of first ANC visit

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Combined retention and treatment failure outcome | Baseline, 3 months postpartum, 6 months postpartum
  Failure will be outcome of a missed visit (>30 days) OR treatment failure (elevated VL>= 200 copies/ml among PWLWH assessed through medical records from baseline to 6 months postpartum.

SECONDARY OUTCOMES:
Depression | Baseline, 3 months postpartum, 6 months postpartum
  Depression score is calculated and severity assessed through a survey utilizing Patient Health Questionnaire Depression Scale (PHQ-9). PHQ-9 score is obtained by adding score for each question (total points). Total score of 0-4 suggests none to minimal depression severity, score of 5-9 mild depression severity, score of 10-14 moderate depression severity, a score of 15-19 moderately severe depression, and a score of 20-27 severe depression.
Psychological Outcome Profiles | Baseline, 3 months postpartum, 6 months postpartum
  Psychological Profile of the study participant is assessed through a survey utilizing Psychological Outcomes Profile scale (PSYCHLOPS). The scale consists of four questions measuring three domains: Problems, Function and Wellbeing. The score is obtained by adding a score for each questions (total points). The maximum score for each question is 5. The maximum PSYCHLOPS score is 20. A higher score indicates a worse outcome.
Fidelity - Content | 6 months postpartum
  The fidelity content measure will be considered reached if 75% or more of observed intervention sessions have all the recommended intervention content fully covered as per the manual Key Points checklist.
Fidelity - Coverage | 6 months postpartum
  Fidelity coverage will be reached if 80% or more of study participants will complete the expected number of sessions.
Feasibility - Recruitment | Enrollment
  The intervention will be considered feasible if the proportion of eligible women able to be recruited into the study per clinic per month equals or exceeds 80% of those eligible for recruitment.
Acceptibility | 6 months postpartum
  The intervention will be considered acceptable if 90% percent or more of intervention participants will rate the intervention completely acceptable. Acceptability will be assessed using items from the Theory-informed questionnaire to assess the acceptability of healthcare interventions. The acceptability outcome indicator will be based on one question from the questionnaire: "How acceptable was the intervention to you? Response options range from completely unacceptable (1) to completely acceptable(5). A higher score means higher acceptability. The intervention will be considered acceptable if 90% or more of intervention participants rate the intervention as completely acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Abuogi, MD, MSc, Principal Investigator — University of Colorado, Denver
Locations (1):
- Kenya Medical Research Institute, Nairobi, Kenya